CLINICAL TRIAL: NCT03266913
Title: Efficacy and Safety of Probiotics in Neonatal Hyperbilirubinemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Mahboobi, Principle Investigator, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4889
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Hyperbilirubinemia, Neonatal
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal | interventions — Probiotics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Active Comparator): Routine phototherapy plus probiotic oral drops at the dose of 10 drops daily
  Interventions: Drug: Probiotic
- No probiotic (No Intervention): Routine phototherapy

INTERVENTIONS:
Drug: Probiotic — Probiotics drop
  Other Names: PediLact
  Arms: Probiotic

SUMMARY:
Neonatal Jaundice occurs in 60% of term infants and 80% of premature infants. Although it is transient, it is associated with high rate of readmission of patients in the first week of infancy. Neonatal jaundice can cause neurological complications and kernicterus. Considering the fact that there have been a lot of studies on probiotic role in management of necrotizing enterocolitis (NEC) and few studies on their role in neonatal jaundice, we carried out this study to determine the efficacy and safety of probiotics in neonatal hyperbilirubinemia in infants hospitalized in children hospital in Bandar Abbas.

ELIGIBILITY:
Inclusion Criteria:

* Between 2 and 28 days old
* Having jaundice
* Gestational age between 35-42 weeks

Exclusion Criteria:

* Less than 2 days or more than 28 days old
* Gestational age out of the range of 35-42 weeks
* Infants whose parents refused to cooperate
* Patients with sepsis and other comorbid conditions

Ages: 2 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-10-01 (Estimated); Study Completion 2017-11-01 (Estimated)

PRIMARY OUTCOMES:
Duration of phototherapy | 6 days
  Duration of phototherapy

SECONDARY OUTCOMES:
Discharge rate | 6 days
  percentage of infants discharged from the hospital at 2nd, 3rd, 4th, and 5th days of admission

CONTACTS AND LOCATIONS:
Overall Officials: Rakhshaneh Goodarzi, M.D, Principal Investigator — Hormozgan University of Medical Sciences
Locations (1):
- Children hospital, Bandar Abbas, Hormozgan, Iran

IPD SHARING:
Plan to Share IPD: Undecided